CLINICAL TRIAL: NCT00113035
Title: Screening Protocol to Evaluate Acid Alpha Glucosidase (GAA) Activity and GAA Gene Mutations in Patients With Late Onset Pompe Disease for Potential Inclusion in Future Clinical Studies With Myozyme (Alglucosidase Alfa)
Brief Title: Screening Protocol to Evaluate Acid Alpha-Glucosidase (GAA) Activity and GAA Gene Mutations in Patients With Late Onset Pompe Disease
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: Sanofi (Industry)
Other Study IDs: AGLU02905
Record Dates: First submitted 2005-06-03; First posted 2005-06-06 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Pompe Disease
Keywords: Glycogen Storage Disease Type II; GSD-II; Pompe Disease; Pompe Disease (Late-Onset); Glycogen Storage Disease Type II (GSD-II); Acid Maltase Deficiency; Glycogenosis 2
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with late onset Pompe Disease

SUMMARY:
Pompe disease (also known as glycogen storage disease type II) is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with Pompe disease, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function. The primary objective of this study is to identify potential candidates for future clinical studies in Pompe disease.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent prior to any study-related procedures being performed
* Clinical presentation consistent with late-onset Pompe disease, or a current clinical diagnosis of late-onset Pompe disease
* Must be greater than or equal to 8 years of age
* Must be able to ambulate (use of assistive devices, such as a walker, cane or crutches, is permitted)

Exclusion Criteria:

* Requires the use of invasive ventilatory support
* Requires the use of noninvasive ventilatory support while awake and in an upright position
* Use of any investigational product within 30 days prior to study enrollment
* Unwillingness to comply with protocol requirements
* Has clinically significant organic disease, unstable medical condition, serious or intercurrent illness
* Is pregnant or lactating
* Has participated in the Prospective Observational Study in Patients with Late-Onset Pompe Disease (AGLU02303, "LOPOS")

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2005-05; Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Tower Hematology/Oncology Medical Group, Beverly Hills, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington University Medical Center, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania